CLINICAL TRIAL: NCT05106283
Title: Comparison of the Effects of Ultrasound-Guided Deep Serratus Anterior Plane Block and Combination of Deep and Superficial Serratus Anterior Plane Block on Postoperative Acute Pain in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Comparison of Deep Serratus Anterior Plane Block and Combination of Deep and Superficial Serratus Anterior Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-2066
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Serratus Anterior Plane Block; Multimodal Analgesia; Thoracic Surgery, Video-Assisted
Keywords: Serratus Anterior Plane Block, Multimodal Analgesia, VATS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Serratus Anterior Plane Block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique beneath the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine will be injected into the area.
  Interventions: Procedure: Deep block and Combined Block
- Deep and Superficial Serratus Anterior Plane Block (Active Comparator): In patients who are planned to have combined deep and superficial serratus anterior plane block, following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique beneath the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 10 ml 0.25% bupivacaine will be injected into the area. Then, with the same needle, will be returned 1-2 cm from the deep serratus anteror area to superficial serratus anteror area above the serratus anterior muscle and will be injected 2 ml normal saline for hydrodissection. Finally 10 ml of 0.25% bupivacaine will be injected for superficial serratus anetrior block into the interfacial area.
  Interventions: Procedure: Deep block and Combined Block

INTERVENTIONS:
Procedure: Deep block and Combined Block — Deep serratus anterior block and combined deep and superficial serratus anterior plane block will be applied to the patients under real-time ultrasound guidance.

SUMMARY:
Video-assisted thoracic surgery (VATS) has become a common procedure in thoracic surgery. Severe postoperative pain may be encountered in patients undergoing VATS. Analgesic methods such as thoracic paravertebral block (TPVB), intercostal block, serratus anterior plane block (SAPB) and erector spina plane block (ESPB) are widely used for VATS. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In recent years, the frequency of application of plane blocks as a component of multimodal analgesia has been increased. ESPB and SAPB are some of them. There are two techniques for SAPB application. In Deep SAPB (DSAPB) application, local anesthetic agent is given under the serratus anterior muscle. In the Superficial SAPB (SSAPB) application, the local anesthetic agent is given above the serratus anterior muscle. Since it is done by entering from the same point in two applications, it is possible to perform these two applications at the same time with a single needle entry. The mechanisms of regional analgesia techniques used after thoracic surgery operations are also different from each other. Therefore, it may be possible to obtain a more effective analgesic effect in patients by combining the mechanism of action of DSAPB and SSAPB , as in the multimodal analgesia method. This study seeks to evaluate the effect of DSAPB and combined DSAPB-SSAPB pain after VATS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective video assisted thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* Chronic opioid or analgesic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 48 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th, 24th and 48th hours after surgery.

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)